CLINICAL TRIAL: NCT05794854
Title: The Assessment of Spot Reduction in Adults Males Following Endurance Training
Brief Title: Spot Reduction in Male Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molde University College (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MUCSR12
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Healthy
Keywords: endurance exercise; subcutaneous tissue utilization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor of dual x-ray absorptiometry results was blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- abdominal aerobic endurance exercise (Experimental): Subjects were combining treadmill running at 70% HRmax (27 minutes) with 4x4minutes (30-40% maximal strength, 1RM) of torso rotation and abdominal crunches (57 minutes), 4 d per wk for 10 weeks
  Interventions: Other: Abdominal aerobic endurance exercise
- Control group (Active Comparator): Subjects performed only treadmill running (45 minutes) at 70% HRmax for 4 d per week for 10 weeks.
  Interventions: Other: Control training intervention

INTERVENTIONS:
Other: Abdominal aerobic endurance exercise — Subjects combined treadmill running at 70% HRmax (27 minutes) with 4x4minutes (30-40% maximal strength, 1RM) of torso rotation and abdominal crunches (57 minutes), 4 days per wk for 10 weeks
  Arms: abdominal aerobic endurance exercise
Other: Control training intervention — Subjects performed treadmill running (45 minutes) at 70% HRmax 4 days per week for 10 weeks
  Arms: Control group

SUMMARY:
Spot reduction, referring to local body fat reduction, pertains to subcutaneous adipose tissue utilization from specific body parts during exercise. Its existence has been keenly debated, although generally accepted not to occur during exercise. However, it is based on not only equivocal data - commonly the training protocol typically applied is based on strength rather than endurance training. The investigators sought to test this assumption by utilizing endurance based exercise controlling for energy expenditure and using dual x-ray absorptiometric measures to assess body composition before and after training.

ELIGIBILITY:
Inclusion Criteria:

* males
* ≥ 30 years old
* classified as overweight (Body mass index ≥ 25 kg ∙ m-2)
* not participating in regular physical training

Exclusion Criteria:

* < 30 years old
* Body mass index < 25 kg ∙ m-2
* participating in regular physical training

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2005-08 (Actual); Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Trunk fat mass change | Change from pre (baseline) to post test (after 10 weeks)
  Fat mass located in trunk (g) measured by dual-energy x-ray absorptiometry

SECONDARY OUTCOMES:
Lower extremity fat mass change | Change from pre (baseline) to post test (after 10 weeks)
  Fat mass located in lower extremities (g) measured by dual-energy x-ray absorptiometry
Upper extremity fat mass change | Change from pre (baseline) to post test (after 10 weeks)
  Fat mass located in upper extremities (g) measured by dual-energy x-ray absorptiometry
Total fat mass change | Change from pre (baseline) to post test (after 10 weeks)
  Total fat mass (g) measured by dual-energy x-ray absorptiometry
Body weight change | Change from pre (baseline) to post test (after 10 weeks)
Body mass index change | Change from pre (baseline) to post test (after 10 weeks)
Waist circumference (cm) change | Change from pre (baseline) to post test (after 10 weeks)
Hip circumference (cm) change | Change from pre (baseline) to post test (after 10 weeks)

OTHER OUTCOMES:
Trunk lean mass change | Change from pre (baseline) to post test (after 10 weeks)
  Lean mass located in trunk (g) measured by dual-energy x-ray absorptiometry
Lower extremity lean mass change | Change from pre (baseline) to post test (after 10 weeks)
  Lean mass located in lower extremities (g) measured by dual-energy x-ray absorptiometry
Upper extremity lean mass change | Change from pre (baseline) to post test (after 10 weeks)
  Lean mass located in upper extremities (g) measured by dual-energy x-ray absorptiometry
Total lean mass change | Change from pre (baseline) to post test (after 10 weeks)
  Total lean mass (g) measured by dual-energy x-ray absorptiometry
Maximal oxygen uptake change | Change from pre (baseline) to post test (after 10 weeks)
  Maximal oxygen uptake by cardiopulmonary indirect calorimetry
Maximal muscle strength change | Change from pre (baseline) to post test (after 10 weeks)
  One-repetition maximum (kg) in torso rotation and abdominal crunch

IPD SHARING:
Plan to Share IPD: No